CLINICAL TRIAL: NCT03914547
Title: Home Video-based Telemedicine to Reduce Hypoglycemia Fear in Parents of Young Children
Acronym: REDCHiP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other); University of Florida (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Susana Patton, Principal Research Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000545; 1R01DK118514-01A1 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REDCHiP intervention arm (Experimental): REDCHiP uses 10- video-based telemedicine sessions to deliver T1D education, behavioral parent training, and problem-solving to enhance parents' knowledge and skills. Sessions last about 45-60 minutes each.
  Interventions: Behavioral: REDCHiP
- Attention Control arm (Active Comparator): ATTN uses 10- video-based telemedicine sessions to deliver general patient education specific to young children. Similar to REDCHiP, all ATTN sessions last 45-60 minutes.
  Interventions: Behavioral: ATTN

INTERVENTIONS:
Behavioral: REDCHiP — REDCHiP includes 10 telehealth sessions. REDCHiP uses a three-pronged approach to reduce parents' FH. It uses T1D education and problem-solving to enhance parents' knowledge and skills. It uses child age-appropriate behavioral parent training to promote parents' skills and confidence in managing disruptive child behaviors and reducing their reliance on hypoglycemia avoidance behaviors. It uses cognitive-behavioral therapy strategies to help parents reduce maladaptive thinking/coping related to hypoglycemia fear.
  Arms: REDCHiP intervention arm
Behavioral: ATTN — Provides a similar attention control. ATTN includes 10 telehealth sessions.
  Arms: Attention Control arm

SUMMARY:
Investigators developed REDCHiP (Reducing Emotional Distress for Childhood Hypoglycemia in Parents), an innovative video-based telemedicine intervention. In the pilot work, investigators found preliminary efficacy for REDCHiP in reducing parental FH, parenting stress, and children's HbA1c. The objective of this clinical trial is to conduct a randomized clinical trial (RCT) comparing REDCHiP to a relevant attention control intervention (ATTN) in families of young children, thereby continuing to establish its efficacy. The proposed R01 aims are: 1) To evaluate whether parents who receive REDCHiP report reductions in FH and parenting stress at post-treatment compared to parents who receive the ATTN; 2) To evaluate whether children of parents who receive REDCHiP have a lower HbA1c and less glycemic variability at post-treatment compared to children of parents who receive ATTN; 3) To examine whether families who receive REDCHiP maintain reductions in FH, parenting stress, and child HbA1c at a 3-month followup compared to families who receive ATTN.

DETAILED DESCRIPTION:
The purpose of this trial is to examine the efficacy of a real-time video-based telemedicine intervention addressing parental fear of hypoglycemia (FH) in families of young children with type 1 diabetes (T1D). Hypoglycemia is a common negative event associated with intensive insulin therapy in children with T1D. Young children with T1D are particularly vulnerable to episodes of hypoglycemia because they tend to be more insulin sensitive, may engage in unpredictable eating and physical activity patterns, and may be less able to recognize and report symptoms. Parents and young children living with T1D quickly learn to fear hypoglycemia because it is uncomfortable, embarrassing, seemingly unpredictable, and potentially dangerous. Indeed, research shows that parents of young children report high rates of moderate to severe FH. Unfortunately, FH leads to two problems: impaired quality of life and compensatory behaviors that raise children's blood glucose levels leading to on-going poor metabolic control (HbA1c) and an increased risk for long-term vascular complications. Responding to a critical need for interventions to treat parental FH in families of young children, investigators developed an innovative video-based telemedicine intervention, called REDCHiP (Reducing Emotional Distress for Childhood Hypoglycemia in Parents). REDCHiP uses cognitive behavioral therapy, T1D education, and behavioral parent training in a 10-session individual and group-based telemedicine program, to reduce parental FH and to teach parents how to change hypoglycemia avoidance behaviors. In the pilot work, investigators found preliminary efficacy for REDCHiP in reducing parental FH, parenting stress, and children's HbA1c. The objective of the proposed R01 is to conduct a randomized clinical trial (RCT) comparing REDCHiP to a relevant attention control intervention (ATTN) in families of young children, thereby continuing to establish its efficacy. The proposed R01 aims are: 1) To evaluate whether parents who receive REDCHiP report reductions in FH and parenting stress at post-treatment compared to parents who receive the ATTN; 2) To evaluate whether children of parents who receive REDCHiP have a lower HbA1c and less glycemic variability at post-treatment compared to children of parents who receive ATTN; 3) To examine whether families who receive REDCHiP maintain reductions in FH, parenting stress, and child HbA1c at a 3-month followup compared to families who receive ATTN. Investigators will recruit 180 families with the goal of retaining at least 144 through the 3-month followup. After informed consent, investigators will randomize parents to either REDCHiP or ATTN and have them complete baseline measures (e.g., parent surveys, child glucose sensing, child/parent accelerometry, and child HbA1c). Then, parents in both groups will participate in 10 video-based telemedicine sessions matched for time and format (group v individual). At post-treatment, parents and children will repeat the baseline assessment; at the 3-month followup, parents will complete surveys and children will undergo glucose sensing and an HbA1c. Primary outcomes of the revised trial are: parents' FH, parenting stress, children's HbA1c levels and children's glycemic variability (measured by percent time above, below and within-range). Secondary measures include child physical activity and sleep, parent sleep, parent depressive symptoms and anxiety, and parent psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* Child age between 2-6.99 years
* Type 1 diabetes diagnosis ≥6 months
* Child is on an intensive insulin regimen (pump or multiple daily injection)

Exclusion Criteria:

* Parents of children on a conventional regimen
* Children who have an allergy or sensitivity to the adhesive and/or skin preparation used for continuous glucose monitoring
* Children with a comorbid chronic condition (e.g., renal disease)
* Parents who do not speak English.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 396 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Child Glycemic Control | change from baseline to post-treatment (week 14)
  Child glycemic control will be measured by change in hemoglobin A1c (HbA1c) NGSP (%) between baseline and post-treatment.
Parents Hypoglycemia Fear | change from baseline to post-treatment (week 14)
  Parental fear will be measured by the Hypoglycemia Fear Survey - Parents of Young Children (HFS-PYC), a 26-item survey with a score range of 26-130. Higher scores indicate a higher fear rating.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - The Children's Mercy Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No
no plan to share individual participant data; de-identified group data may be available to qualified researchers upon request to the principal investigator

REFERENCES:
- [Derived] Patton SR, McConville A, Marker AM, Monzon AD, Driscoll KA, Clements MA. Reducing Emotional Distress for Childhood Hypoglycemia in Parents (REDCHiP): Protocol for a Randomized Clinical Trial to Test a Video-Based Telehealth Intervention. JMIR Res Protoc. 2020 Aug 18;9(8):e17877. doi: 10.2196/17877. PMID 32808936